CLINICAL TRIAL: NCT02194335
Title: A Double-blind (Within Dose Groups), Randomised, Placebo-controlled Single Increasing Dose Safety, Tolerability and Pharmacokinetics Study (Parallel Groups) in Healthy Male and Female Volunteers After Oral Administration of BIBN 4096 BS Drinking Solution (Dosage: 20 - 200 mg)
Brief Title: Safety, Tolerability and Pharmacokinetics of Increasing Doses of BIBN 4096 BS in Healthy Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1149.34
Record Dates: First submitted 2014-07-17; First posted 2014-07-18 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-07

CONDITIONS: Healthy

ARMS (2):
- BIBN 4096 BS - in single rising doses (Experimental)
  Interventions: Drug: BIBN 4096 BS - in single rising doses
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIBN 4096 BS - in single rising doses
  Arms: BIBN 4096 BS - in single rising doses
Drug: Placebo
  Arms: Placebo

SUMMARY:
The objective of the present study was to obtain information about safety, tolerability and pharmacokinetics of BIBN 4096 BS after oral administration of increasing doses in healthy male and female volunteers. With respect to pharmacokinetics, it was of particular importance to investigate whether therapeutic plasma levels (for treatment of migraine) could have been achieved by oral administration of a BIBN 4096 BS formulation.

ELIGIBILITY:
Inclusion Criteria:

* Participants should be healthy males and females
* Age range from 21 to 50 years
* Broca Index: within +- 20% of their normal weight
* Subsequently each subject will have his medical history taken and will receive a complete medical examination (incl. blood pressure and pulse rate measurements) as well as a 12-lead Electrocardiogram (ECG). Hematopoietic, hepatic and renal function test will be carried out in the laboratory. The subjects will fast for 12 hours before collection of specimens for all laboratory evaluations. The above mentioned examinations will be performed within 14 days before the first administration of the test substance. In accordance with Good Clinical Practice (GCP) and local legislation all volunteers will have given their written informed consent prior to admission to the study

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Diseases of the central nervous system (such as epilepsy) or with psychiatric disorders or neurological disorders
* History of orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (>24 hours) within at least one month or less than ten half-lives of the respective drug before enrolment in the study (exclusion: substitution therapy regarding thyroid gland and/or ovaries)
* Use of any drugs which might influence the results of the trial (within one week prior to administration or during the trial)
* Participation in another study with an investigational drug within two months prior to administration or during the trial
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking on study days
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation (>= 100 ml) within four weeks prior to administration or during the trial
* Excessive physical activities (within the last week before the study)
* Any laboratory value outside the reference range of clinical relevance

For female subjects:

* Pregnancy
* Positive pregnancy test
* No adequate contraception e.g. oral contraceptives, sterilization, intrauterine pessary (IUP)
* Inability to maintain this adequate contraception during the whole study period
* Lactation period

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2000-10; Primary Completion 2000-12 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | up to 24 days
Number of patients with abnormal changes in laboratory parameters | up to 8 days after drug administration
Number of patients with clinically significant changes in vital signs (blood pressure, pulse rate) | up to 8 days after drug administration
Number of patients with clinically significant changes in 12-lead Electrocardiogram (ECG) | up to 8 days after drug administration

SECONDARY OUTCOMES:
AUC0-∞ (Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 24 hours after drug administration
Cmax (Maximum measured concentration of the analyte in plasma) | up to 24 hours after drug administration
tmax (Time from dosing to the maximum concentration of the analyte in plasma) | up to 24 hours after drug administration
CL/F (Apparent clearance of the analyte in plasma following extravascular administration) | up to 24 hours after drug administration
t½ (Terminal half-life of the analyte in plasma) | up to 24 hours after drug administration
MRTtot (Total mean residence time of the analyte in plasma) | up to 24 hours after drug administration
Vz/F (Apparent volume of distribution of the analyte during the terminal phase) | up to 24 hours after drug administration
AUC0-tz (Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point) | up to 24 hours after drug administration
Terminal rate constant in plasma | up to 24 hours after drug administration